CLINICAL TRIAL: NCT06736704
Title: A Phase 1/2, Open-Label Dose Escalation and Expansion Study of SNV4818 as Monotherapy or in Combination With Other Anticancer Agents in Participants With Advanced Solid Tumors
Brief Title: SNV4818 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pikavation Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNV4818-101
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Fulvestrant; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SNV4818 Monotherapy (Experimental): Participants will receive oral, daily doses of SNV4818 as a single agent as part of either dose escalation or dose expansion cohorts. The SNV4818 dose level participants receive will depend upon the study part to which they are assigned. Dose escalation participants will be assigned to small cohorts of ascending SNV4818 dose levels. Dose expansion participants will receive one of the SNV4818 dose levels recommended for further evaluation.
  Interventions: Drug: SNV4818
- SNV4818+Fulvestrant Combination (Experimental): Participants will receive oral, daily doses of SNV4818 in combination with a standard dose of Fulvestrant as part of either dose escalation or dose expansion cohorts.. The SNV4818 dose level participants receive will depend upon the study part to which they are assigned. Dose escalation participants will be assigned to small cohorts of ascending SNV4818 dose levels. Dose expansion participants will receive one of the SNV4818 dose levels recommended for further evaluation.
  Interventions: Drug: SNV4818; Drug: Fulvestrant
- SNV4818+Palbociclib+Fulvestrant Combination (Experimental): Participants will receive oral, daily doses of SNV4818 in combination with a standard doses of Palbociclib and Fulvestrant as part of either dose escalation or dose expansion cohorts.. The SNV4818 dose level participants receive will depend upon the study part to which they are assigned. Dose escalation participants will be assigned to small cohorts of ascending SNV4818 dose levels. Dose expansion participants will receive one of the SNV4818 dose levels recommended for further evaluation.
  Interventions: Drug: SNV4818; Drug: Fulvestrant; Drug: Palbociclib

INTERVENTIONS:
Drug: SNV4818 — SNV4818 is a tablet taken orally. Dose and frequency are dependent upon treatment arm.
Drug: Fulvestrant — Fulvestrant is administered via an intramuscular injection. It will be given at a dose of 500 mg (2-250 mg/5 mL injections)
  Other Names: Faslodex
  Arms: SNV4818+Fulvestrant Combination; SNV4818+Palbociclib+Fulvestrant Combination
Drug: Palbociclib — Palbociclib tablets will be administered by mouth on days 1-21 of a 28 day cycle. The Palbociclib starting dose will be 125 mg once-daily
  Other Names: Ibrance
  Arms: SNV4818+Palbociclib+Fulvestrant Combination

SUMMARY:
This study is testing a new medicine, SNV4818, for people with advanced cancers. The researchers want to find out if SNV4818 is safe, well-tolerated, and effective in treating solid tumors. They are investigating different doses in order to find the safest and most effective one.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic solid tumor with an activating PIK3CA mutation.
* Refractory to or intolerant of available therapies
* Disease measurable by RECIST 1.1 criteria, or disease evaluable by clinically relevant tumor biomarkers in blood.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Diagnosis of a primary CNS malignancy
* Active brain metastases or carcinomatous meningitis
* Type 1 diabetes mellitus or uncontrolled type 2 diabetes mellitus
* Inadequate organ function
* Clinically significant ECG abnormalities, including QTcF ≥ 470 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) | First 28 days of study treatment
  -Number of participants experiencing protocol-defined DLTs (Part 1A and 2A only)
Treatment Emergent Adverse Events (TEAEs) | From first SNV4818 dose through approximately 30 days following the last SNV4818 dose
  Incidence and frequency of TEAEs

SECONDARY OUTCOMES:
Maximum observed plasma concentration of SNV4818 | After 4 weeks (1 cycle) of study treatment
  Cmax
Time to reach the maximum observed plasma concentration of SNV4818 | After 4 weeks (1 cycle) of study treatment
  Tmax
Area Under Plasma Concentration (AUC) Time Curve of SNV4818 | After 4 weeks (1 cycle) of study treatment
  AUC0-t
Half-life of SNV4818 | After 4 weeks (1 cycle) of study treatment
  t1/2
Area Under Plasma Concentration (AUC) Time Curve of SNV4818 extrapolated to infinity | After 1 day of study treatment
  AUC0-infinity
Apparent oral clearance of SNV4818 | After 4 weeks (1 cycle) of study treatment
  CL/F
Apparent volume of distribution of SNV4818 | After 4 weeks (1 cycle) of study treatment
  Vz/F
Overall response rate (ORR) | After 8 weeks on study treatment
  The proportion of participants who achieve a best overall response (BOR) of complete response (CR) or partial response (PR), based on RECIST 1.1 criteria
Disease control rate (DCR) | After 8 weeks on study treatment
  The proportion of participants who have a best overall response (BOR) of stable disease (SD) or better
Duration of response (DOR) | Up to approximately 2 years
  The time interval between an assessment of partial response (PR) or better and disease progression or death due to any cause.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Thomas Jefferson University-Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Scientia Clinical Research, Randwick, New South Wales
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - University Health Network, Princess Margaret Cancer Centre, Toronto, Ontario